CLINICAL TRIAL: NCT03931200
Title: Real World Demographic and Clinical Characteristics, Treatment Patterns and Clinical Outcomes of Heart Failure Patients in China: a Retrospective Non-Interventional Nationwide Study
Brief Title: Demographic and Clinical Characteristics, Treatment Patterns and Clinical Outcomes of Heart Failure Patients in China
Status: Completed | Type: Observational
Sponsor: China Cardiovascular Association (Other)
Responsible Party: Sponsor
Other Study IDs: GUSU19002
Record Dates: First submitted 2019-04-15; First posted 2019-04-30 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, multicenter, retrospective study assessing demographic characteristics, clinical characteristics, management and outcome of patients with a HF (heart failure) diagnosis utilizing real world data derived from HF Center Database. This database collects the data of HF from patients hospitalized between March 2010 to Dec 2018 in more than 300 hospitals across China.

DETAILED DESCRIPTION:
Research question and objectives Primary objective

* Describe the demographic and clinical characteristics of HF patients at HF index hospitalization admission Secondary objective
* Assess the HF diagnosis and evaluation patterns and treatment patterns during index hospitalization and after discharge compare with guideline (2018 China HF Guideline) recommendations
* Describe the demographic characteristics, clinical characteristics, diagnostic pattern, treatment pattern of HF patients stratified by LVEF (left ventricular ejection fraction) and region Exploratory objectives Describe the demographic and clinical characteristics, sac/val start dose and titration pattern among chronic HF patients prescribed sac/val

Study design This is a non-interventional, multicenter, retrospective study assessing demographic characteristics, clinical characteristics, management and outcome of patients with a HF diagnosis utilizing real world data derived from HF Center Database. This database collects the data of HF from patients hospitalized between March 2010 to Dec 2018 in more than 300 hospitals across China.

Setting and study population This study will include the data from all patients who were enrolled in the HF Center database. The study population consists of adult inhospital patients (18+ years) being diagnosed with HF at discharge.

Inclusion criteria

* Aged 18 years and older
* Patients with confirmed diagnosis of HF
* Diagnosis is made by the treating physicians according to local practices and their clinical judgement Exclusion criteria Concomitant participation in a clinical study with any investigational treatment during the index hospitalization

Variables

Collection at index hospitalization:

Demography Comorbidities and Medical History Patient presentation at admission (including signs and symptoms) Vital Status In-hospital evaluation tests (laboratories, function tests, etc) Medication at discharge

Collection at follow-up (1 month, 3months and 1year):

Vital status Evaluation tests (laboratories, function tests, etc) Medication at follow-up Clinical outcomes (mortality and re-hospitalization events where feasible)

Data sources The data from this study will be retrieved from the HF Center database provided by CHH (China Heart House). All data were collected from more than 300 collaborative hospitals of China, including approximately 60,000 patients of HF. The information was collected during index hospitalization, 1 month, 3 months, 1 year after discharge by trained coordinators using a standardized case report form, entered into the HF Center database.

Study size This study will be conducted based on existing database and no formal sample size calculation is necessary for this type of descriptive retrospective observational research. In HF Center database, there is around 60,000 patients in total planned to be analyzed in this study.

Data analysis Descriptive data analyses will be focus on: (1) Continuous variables: mean, standard error, median, first quartile, third quartile, ranges for continuous variables; (2) Categorical variables: frequencies, and percentages for categorical variables. Summaries will be presented together with estimates and corresponding 95% confidence intervals (CI) as appropriate.

For the endpoints that stratified by LVEF and region, differences will be assessed by the p-values of corresponding tests. Categorical variables will be compared using chi-square tests; continuous variables will be compared using unequal variance two-sample t-test; for continuous variables with skewed data Mann-Whitney U test will be used, or Wilcoxon signed-rank test in case of paired data. 95% confidence intervals (CIs) and two tailed p-value will be reported for the parameter estimated in the multivariable models.

The number and proportion of patients with missing data will be presented. Detailed description will be provided in the SAP (Statistical Analysis Plan).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Patients with confirmed diagnosis of HF
* Diagnosis is made by the treating physicians according to local practices and their clinical judgement

Exclusion Criteria:

• Concomitant participation in any/a clinical trial with any investigational treatment during the index hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The demographic and clinical characteristics were collected from patients' medical records during their in-patients treatment period, and the follow-up data were collected from face-to-face interview at outpatient clinics or phone interview after discharge.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Patients' demographics at index hospitalization admission. | 1 years
  Patients' demographics at index hospitalization admission.
Patients' medical history at index hospitalization admission. | 1 years
  Patients' medical history at index hospitalization admission.
Patients' comorbidities (i.e. diabetes, renal insufficiency, chronic obstructive pulmonary disease, anemia, obesity, hypertension) at index hospitalization admission. | 1 years
  Patients' comorbidities (i.e. diabetes, renal insufficiency, chronic obstructive pulmonary disease, anemia, obesity, hypertension) at index hospitalization admission.

SECONDARY OUTCOMES:
The percentage of patients who received the guideline (2018 China HF Guideline) recommended tests during the indexed hospitalization. | 1 years
  The percentage of patients who received the guideline (2018 China HF Guideline) recommended tests (i.e. echocardiography, electrocardiogram, brain natriuretic peptide (BNP)/n-terminal pro-brain natriuretic Peptide (NT-proBNP)) during the indexed hospitalization.
The percentage of HF patients who received the guideline (2018 China HF Guideline) recommended HFrEF (Hear failure with reduced ejection fraction) pharmacological and device treatments (i.e. ICD, CRT) at the discharge of the index hospitalization. | 1 years
  The percentage of HF patients who received the guideline (2018 China HF Guideline) recommended HFrEF pharmacological (i.e. Angiotensin-converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), ARNI, β-blockers, aldosterone antagonists, diuretics) and device treatments (i.e. ICD, CRT) at the discharge of the index hospitalization.
The percentage of HF patients adherent to guideline. | 1 years
  The percentage of HF patients adherent to guideline (2018 China HF Guideline) recommended HFrEF pharmacological treatments including ACEIs, ARBs, β-blockers, aldosterone antagonists and diuretics at 1 month, 3 months and 1 year after discharge from the indexed hospitalization.
Follow-up rate at 1month, 3 months and 1 year after discharge from indexed hospitalization. | 1 years
  Follow-up rate at 1month, 3 months and 1 year after discharge from indexed hospitalization.
In-hospital mortality rate at 1month, 3 months and 1 year after discharge from indexed hospitalization. | 1 years
  In-hospital mortality rate at 1month, 3 months and 1 year after discharge from indexed hospitalization.
Re-hospitalization rate at 1month, 3 months and 1 year after discharge from indexed hospitalization. | 1 years
  Re-hospitalization rate at 1month, 3 months and 1 year after discharge from indexed hospitalization.
Demographic characteristics among HF patients stratified by LVEF (<40%/40-49%/≥50%). | 1 years
  Demographic characteristics among HF patients stratified by LVEF (<40%/40-49%/≥50%).
Medical history among HF patients stratified by LVEF (<40%/40-49%/≥50%). | 1 years
  Medical history among HF patients stratified by LVEF (<40%/40-49%/≥50%).
Diagnostic pattern among HF patients stratified by LVEF (<40%/40-49%/≥50%). | 1 years
  Diagnostic pattern among HF patients stratified by LVEF (<40%/40-49%/≥50%).
Treatment pattern among HF patients stratified by LVEF (<40%/40-49%/≥50%). | 1 years
  Treatment pattern among HF patients stratified by LVEF (<40%/40-49%/≥50%).
Outcomes among HF patients stratified by LVEF (<40%/40-49%/≥50%). | 1 years
  Outcomes among HF patients stratified by LVEF (<40%/40-49%/≥50%).
Demographic characteristics comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China. | 1 years
  Demographic characteristics comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China.
Medical history comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China. | 1 years
  Medical history comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China.
Diagnostic pattern comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China. | 1 years
  Diagnostic pattern comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China.
Treatment pattern comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China. | 1 years
  Treatment pattern comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China.
Outcomes comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China. | 1 years
  Outcomes comparing HF patients in Shanghai vs the whole of China and Shanghai vs the rest of China.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing hospital, Beijing, Beijing Municipality

REFERENCES:
- [Background] Gu DF, Huang GY, He J, et al (2003). Investigation of prevalence and distributing feature of chronic heart failure in Chinese adult population. Chin J Cardiol, Vol.31,pp.3-6.
- [Background] Huang J, Yin H, Zhang M, Ni Q, Xuan J. Understanding the economic burden of heart failure in China: impact on disease management and resource utilization. J Med Econ. 2017 May;20(5):549-553. doi: 10.1080/13696998.2017.1297309. Epub 2017 Mar 12. PMID 28286996
- [Background] Zhang Y, Zhang J, Butler J, Yang X, Xie P, Guo D, Wei T, Yu J, Wu Z, Gao Y, Han X, Zhang X, Wen S, Anker SD, Filippatos G, Fonarow GC, Gan T, Zhang R; China-HF Investigators. Contemporary Epidemiology, Management, and Outcomes of Patients Hospitalized for Heart Failure in China: Results From the China Heart Failure (China-HF) Registry. J Card Fail. 2017 Dec;23(12):868-875. doi: 10.1016/j.cardfail.2017.09.014. Epub 2017 Oct 10. PMID 29029965
- [Background] ISPE. Guidelines for good pharmacoepidemiology practices (GPP). Pharmacoepidemiol Drug Saf. 2008 Feb;17(2):200-8. doi: 10.1002/pds.1471. No abstract available. PMID 17868186